CLINICAL TRIAL: NCT06972641
Title: A Prospective, Multicenter Umbrella Study Based on Molecular Genetics to Guide the Efficacy and Safety of Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation for Acute Myeloid Leukemia/Myelodysplastic Syndrome
Brief Title: Molecular Genetics Guide the Maintenance Therapy After Allogeneic Hematopoietic Stem Cell Transplantation
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, Hu Xiaoxia, Prof, Ruijin Hospital
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20250404
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-18 (Actual); Status verified 2025-04

CONDITIONS: AML; MDS
MeSH Terms: interventions — Decitabine; Sorafenib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- ARM3: KIT mutation (Experimental): Initial bone marrow gene II sequencing showed KIT mutations (loci: D816, N822, exon 8, VAF ≥2%, excluding germline mutations); no TP53 mutations, AML/MR, FLT3-ITD;
  Interventions: Drug: Avastinib
- ARM2: FLT3-ITD mutation (Experimental): Initial bone marrow gene II sequencing showed FLT3-ITD mutation with or without NPM1 mutation, no TP53 mutation, and no AML/MR.
  Interventions: Drug: Sorafenib (BAY-43-9006)，giritinib
- ARM1 TP53 mutation and/or AML-MR (Experimental): TP53 mutation (VAF ≥ 2%, excluding germline mutations), and/or AML-MR (SRSF2, SF3B1, U2AF1, ZRSR2, ASXL1, EZH2, BCOR, STAG2) by second-generation sequencing of the initial bone marrow gene.
  Interventions: Drug: Decitabine
- ARM4: Other mutations/fusions (Experimental): MDS in the intermediate/high/very high risk group as assessed by IPSS-M or AML in the intermediate/high risk group as assessed by ELN2022 without ARM1, 2, or 3 related mutations/fusions;
  Interventions: Drug: Venetoclax;Selenisol

INTERVENTIONS:
Drug: Decitabine — Decitabine 3.5 mg/m2 1-5d for 28 days for 6 cycles of dosing
  Arms: ARM1 TP53 mutation and/or AML-MR
Drug: Sorafenib (BAY-43-9006)，giritinib — Sorafenib 0.2g 2/day or giritinib 40mg 2/day orally for 2 years
  Arms: ARM2: FLT3-ITD mutation
Drug: Avastinib — 100 mg 1/day
  Arms: ARM3: KIT mutation
Drug: Venetoclax;Selenisol — Vinaclat: 50-100mg 1/day orally, d1-14 1/day per month (adjust drug dosage based on blood levels), 28-day cycle; Selenisol: 20mg qw orally (weeks 1 and 2), 28-day cycle If the above treatment is not tolerated, adjust the regimen to decitabine 3.5 mg/m2 1-5 d; 28 days as a cycle of 6 cycles of medication; Vinaclat: 50-100 mg 1/day orally, d1-14 1/day per month orally (adjust the dose of the drug according to the blood concentration), 28 days as a cycle of medication
  Arms: ARM4: Other mutations/fusions

SUMMARY:
This study is a prospective, multicenter, open-label umbrella clinical study planned to enroll 126 subjects with acute myeloid leukemia/myelodysplastic syndromes undergoing allogeneic hematopoietic stem cell transplantation. Subjects eligible for enrollment were grouped based on the results of the initial myeloid genomic second-generation sequencing, and were given different regimens of maintenance therapy, with the aim of evaluating the efficacy and safety of the maintenance regimen.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, open-label, umbrella study designed to evaluate the efficacy and safety of mutation-based guided post-transplantation maintenance therapy in post-transplantation patients . The study will include allogeneic hematopoietic stem cell transplantation patients who meet the enrollment criteria, applying myeloid gene second-generation sequencing data to classify the patients into four subgroups and set the corresponding treatment arms according to the underlying molecular characteristics of the different subgroups, which will be treated with cerinisol in combination with vinaiquelat, FLT3 inhibitors, avastinib, and decitabine, respectively. Maintenance therapy was initiated 60-90 days post-transplant and continued for a total of 2 years. The study is divided into a screening period (screening is initiated 30-60 days post-transplant) and a treatment follow-up period (after screening, subjects are scheduled for treatment. Maintenance therapy is initiated 60-90 days post-transplantation with follow-up monitoring). Until one of the following occurs: disease progression, toxicity intolerance, or other reasons as specified in the protocol. Subjects who end treatment enter the follow-up period for safety or survival follow-up.

ELIGIBILITY:
Inclusion Criteria:

* 1) Age 14-75 years and gender; (2) Initial diagnosis, pre-transplant myelogenetic second-generation sequencing data refinement; 3)ARM1: TP53 mutation (VAF ≥ 2%, excluding germline mutations), and/or AML-MR (SRSF2, SF3B1, U2AF1, ZRSR2, ASXL1, EZH2, BCOR, STAG2) by second-generation sequencing of the initial bone marrow gene; ARM2 Initial bone marrow gene II sequencing showed FLT3-ITD mutation with or without NPM1 mutation, no TP53 mutation, and no AML/MR. ARM3 Initial bone marrow gene II sequencing showed KIT mutations (loci: D816, N822, exon 8, VAF ≥2%, excluding germline mutations); no TP53 mutations, AML/MR, FLT3-ITD; ARM4 MDS in the intermediate/high/very high risk group as assessed by IPSS-M or AML in the intermediate/high risk group as assessed by ELN2022 without ARM1, 2, or 3 related mutations/fusions; 4) Subjects receive their first allogeneic hematopoietic stem cell transplantation within 30-60 days and STR-PCR shows complete donor chimerism; 5) Evaluation of the primary disease prior to maintenance therapy as complete remission and negative bone marrow flow MRD; 6) No active infection and no acute graft-versus-host disease requiring systemic treatment 7) Have appropriate organ function and laboratory results within 7 days prior to the start of treatment need to meet the following criteria:
* Aspartate aminotransferase (AST) ≤ 3 times ULN (upper limit of normal, ULN);
* Alanine aminotransferase (ALT) ≤ 3x ULN;
* Total serum bilirubin ≤ 1.5 times the upper limit of normal ULN unless the patient has documented Gilbert's syndrome; patients with Gilbert's syndrome with bilirubin ≤ 3.0 times the upper limit of normal and direct bilirubin ≤ 1.5 times the upper limit of normal may be included;
* Hemoglobin ≥ 70 g/L (had not received a red blood cell transfusion within 1 week prior to administration); Absolute neutrophil count (ANC) ≥ 0.8 x 10^9/L (had not received long-acting colony-stimulating factor (LACSF) within 1 week prior to administration and short-acting colony-stimulating factor (SACSF) within 3 days prior to administration); and Platelet count ≥ 20 x 10^9/L (1 week prior to administration) have not received a platelet transfusion);
* Serum creatinine ≤ 1.5 times ULN or creatinine clearance ≥ 60 mL/min;
* Coagulation function: International Normalized Ratio (INR) ≤1.5×ULN, Activated Partial Thromboplastin Time (APTT) ≤1.5×ULN;
* Left ventricular ejection fraction (LVEF) ≥45%; 8) Women of childbearing potential must have a negative serum pregnancy study within 7 days prior to the first dose. Female subjects of childbearing potential and male subjects whose partner is a woman of childbearing potential must agree to use a highly effective method of contraception from the time of signing the informed consent form until 180 days after the last dose of study drug is given (9) Voluntarily signing the informed consent, understanding and complying with the requirements of the study, good compliance, and cooperating with the follow-up visits.

Exclusion Criteria:

Patients were not enrolled if they met any of the following criteria:

1. Bone marrow or peripheral blood MRD changes from negative to positive;
2. Presence of acute or chronic GVHD, active infection requiring systemic immunosuppressive therapy prior to maintenance therapy;
3. Have clinically significant active cardiovascular disease such as uncontrolled arrhythmias, uncontrolled hypertension, congestive heart failure, any grade 3 or 4 heart disease as determined by the New York Heart Association (NYHA) functional class, or a history of myocardial infarction within the 6 months prior to screening;
4. Other serious medical conditions that may limit the patient's participation in this trial (e.g., uncontrolled diabetes, active autoimmune disease, etc.);
5. Known human immunodeficiency virus (HIV) infection, or chronic infection with hepatitis B virus (HBsAg-positive) or hepatitis C virus (anti-HCV-positive) that is uncontrolled by drugs;
6. Patients with neurological or psychiatric disorders;
7. Those who are unable to understand or comply with the study protocol or are unable to sign the informed consent form;
8. The researcher does not consider it appropriate to participate in this study.

Ages: 14 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 126 (Estimated)
Dates: Start 2025-06-10 (Estimated); Primary Completion 2030-03-31 (Estimated); Study Completion 2030-03-31 (Estimated)

PRIMARY OUTCOMES:
EFS | 2 years after transplantation
  Event-free survival

SECONDARY OUTCOMES:
OS | 2 years after transplantation
  Overall survival

CONTACTS AND LOCATIONS:
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared publicly to protect participant confidentiality, as specified in the study's informed consent documents. Even de-identified data may contain sensitive information that could risk re-identification. Aggregate results will be published, and requests for limited data access may be considered after completion of secondary analyses through a formal proposal process approved by the ethics committee.